CLINICAL TRIAL: NCT04518540
Title: Randomized, Parallel Safety and Efficacy Study of Lipoic Acid in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Explore Neuroprotective Effect of Lipoic Acid in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-375
Record Dates: First submitted 2020-08-05; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcomes assessors who do all the scales are concealed of group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lipoic acid group (Experimental): The patients will take lipoic acid by intravenous. At the same time, the patients will take take riluzole tablets orally everyday.
  Interventions: Drug: lipoic acid group
- control group (Experimental): The patients will take riluzole tablets orally everyday.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: lipoic acid group — The patients will take lipoic acid for 6 course, the first course of treatment is 14 days with 14 days of rest, and the following course is the first for 10 days, with 14 days interval.The patients will use 600mg domestic lipoic acid in 250ml normal saline by intravenous, once a day.
  At the same time, the patients will take domestic riluzole tablets 50mg orally, twice a day.
  Arms: lipoic acid group
Drug: control group — The patients will take domestic riluzole tablets 50mg orally, twice a day.
  Arms: control group

SUMMARY:
In this proposed study, the investigators will evaluate the safety and efficacy of lipoic acid in treatment of Amyotrophic lateral sclerosis (ALS). The study will recruit 150 AD patients, and then these patients will be randomized to lipoic acid group or control group (75 patients per arm) for 6 courses for about 5 months. Clinical assessment will be done at screen/baseline, 3th course and 6th course. The specific aims are to compare lipoic acid versus control on: motor function and disease progression. During the study period, clinical effect index will be recorded, including bulbar function, motor function, respiratory function, and safety index including blood and urine routine, liver and kidney function, coagulation function.

DETAILED DESCRIPTION:
In this proposed study, the investigators will evaluate the safety and efficacy of Lipoic acid in treatment of ALS. The study will recruit 150 ALS patients, then these patients will be randomized to lipoic acid group or control group (75 patients per arm) for 6 courses for about 5 months. Clinical efficacy and safety assessment will be done at screen/baseline, 3th course and 6th course. The specific aims are to compare lipoic acid versus placebo on: (1) Lipoic acid could improve the motor function, delay the disease progression and extend survival time in patients with ALS, measured by the ALSFRS-R Scale, ROADS Scale, upper motor neuron Scale, Muscle strength Scale and Electromyography; (2) Lung function will be collected to prove the hypothesis lipoic acid may help respiratory function. (3) Safety index including blood and urine routine, liver and kidney function, coagulation index will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 20 to 75 (including 20 and 75 years old), regardless of ethnic group or gender;
2. The subjects should meet the diagnostic criteria for ALS by El Escorial revised criteria: "Definite ALS", "Probable ALS" and "Probable, laboratory-supported ALS".
3. ALS Functional Rating Scale-Revised (ALSFRS-R 12 items) each item score ≥2 points;
4. The onset (the symptoms of limbs weakness, muscle atrophy or bulbar involvement ) of the disease is less than 2 years
5. Baseline breath function: Forced Vital Capacity≥70% .
6. Disease Progression Rate FS=(48- ALSFRS-R at "time of diagnosis")/duration from onset to diagnosis (month), progression rate FS≤1;

Exclusion Criteria:

1. Combined with one of cerebrovascular disease, spinal cord disease, spinal muscular atrophy, juvenile myoatrophy of distal upper extremity, multifocal motor neuropathy, Kennedy disease, epilepsy, etc;
2. Severe renal insufficiency: creatinine clearance rate <30 mL/min (Cockcroft-Gault formula, urea nitrogen and (or) blood creatinine> 1.5 times the upper limit of normal, or other known severe renal insufficiency diseases;
3. Severe liver damage: ALT, AST> 3 times the upper limit of normal, or other known liver diseases such as acute and chronic hepatitis, cirrhosis, etc.;
4. Obvious tachycardia or bradycardia; patients with acute myocardial infarction or interventional therapy in the past 6 months (patients with grade III-IV according to NYHA classification);
5. Combined with malignant tumor, blood, digestion or other serious diseases;
6. Female patients during pregnancy and lactation;
7. Participated in other clinical trials within 30 days before randomization, or are participating in other clinical trials;

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
change of Amyotrophic lateral sclerosis Function Rate Scale-Revised (ALSFRS-R) | change from baseline to 11th week& 21th week
  The Amyotrophic lateral sclerosis Function Rate Scale-Revised (ALSFRS-R) will be performed to test the motor function of patients at the enrollment, 3th course and 6th course . The score ranges from 0 to 48#and higher scores represent a better motor function.

SECONDARY OUTCOMES:
change of Rasch Overall ALS Disability Scale (ROADS) | change from baseline to 11th week& 21th week
  Rasch Overall ALS Disability Scale (ROADS) will be performed to test the motor function of patients at the enrollment, 3th course and 6th course . The score ranges from 0 to 56#and higher scores represent a better motor function.
change of Upper motor neuron scale (UMNS) | change from baseline to 11th week& 21th week
  Upper motor neuron scale(UMNS) will be performed to test the motor function of patients at the enrollment, 3th course and 6th course . The score ranges from 0 to 33.
change of Muscle strength scale | change from baseline to 11th week& 21th week
  Muscle strength scale will be performed to test the muscle strength of patients at the enrollment, 3th course and 6th course. Higher scores represent a better muscle strength.
change of Pulmonary Forced Vital Capacity (PFVC) | change from baseline to 11th week& 21th week
  Pulmonary Forced Vital Capacity (PFVC) will be performed to test the breath function of patients at the enrollment, 3th course and 6th course. Higher scores represent a better pulmonary function.
change of Motor Neuron Disease Electromyography | change from baseline EMG to 21th week
  Motor Neuron Disease Electromyography will be performed to test the electrical activity of muscles of patients at the enrollment, 3th course and 6th course .

OTHER OUTCOMES:
Endpoint events occur rate | at 21th week
  Endpoint events occur rate, including death, tracheotomy, invasive ventilator assisted ventilation or continuous noninvasive ventilator assisted ventilation (use time ≥22 hours per day, duration ≥10 days);
percentage of adverse drug reaction | At the baseline, 11th week and 21th week
  Check the percentage of adverse drug reactions in blood routine, blood biochemistry, and urine routine

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China